CLINICAL TRIAL: NCT03049137
Title: Evaluation of Computer-Guided Versus Conventional Simultaneous Implant Placement With Ridge Augmentation Using an Autogenous Bone Ring Graft With PRF on Patient's Esthetic Satisfaction
Brief Title: Computer Guided Versus Conventional Augmentation Using Bone Ring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Younis, Dentist at Ministry Of Health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoBRG-PRF
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Surgery, Computer-Assisted; Transplantation, Autologous; Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double Blind (Subject, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Guided Stent Augmentation (Experimental): Patients with defective maxillary anterior alveolar ridges requiring implant insertion will have simultaneous implant placement with ridge augmentation using autogenous bone ring graft covering them with Platelet-rich fibrin (PRF) using computer guided stent.
  Interventions: Procedure: Computer Guided Stent Augmentation; Drug: Platelet-rich fibrin (PRF); Device: implant
- Free Hand Augmentation (Active Comparator): Patients with defective maxillary anterior alveolar ridges requiring implant insertion will have simultaneous implant placement with ridge augmentation using Free hand simultaneous implant placement with ridge augmentation and covering them with Platelet-rich fibrin (PRF).
  Interventions: Procedure: Free Hand Augmentation; Drug: Platelet-rich fibrin (PRF); Device: implant

INTERVENTIONS:
Procedure: Computer Guided Stent Augmentation — Defective alveolar ridge is to be replaced by simultaneous implant placement with ring graft augmentation (Trephine Drill to obtain the ring graft autogenous bone) using computer guided stent and covered with Platelet-rich fibrin (PRF), by using venous blood from the patient, a centrifuge will be used to obtain the top layer after centrifuging blood at 3000 Revolution Per Minute (RPM) for 10 minutes.
  Other Names: Computer Guided Surgery; Autograft
  Arms: Computer Guided Stent Augmentation
Procedure: Free Hand Augmentation — Defective alveolar ridge is to be replaced by Free Hand simultaneous implant placement with ring graft augmentation (Trephine Drill to obtain the ring graft autogenous bone) and covered with Platelet-rich fibrin (PRF), by using venous blood from the patient, a centrifuge will be used to obtain the top layer after centrifuging blood at 3000 RPM for 10 minutes.
  Other Names: Autograft
  Arms: Free Hand Augmentation
Drug: Platelet-rich fibrin (PRF)
Device: implant

SUMMARY:
Using bone ring grafts with simultaneous implant placement after three-dimensional augmentation of severely defective bone ridges using computer-guided surgical templates. The study compares accuracy effectiveness by mimics software

DETAILED DESCRIPTION:
To study the effectiveness of computer guided surgical stents in ridge augmentation with implant insertion compared with free hand augmentation

-Population/Intervention/Comparator/Outcome (PICO)-

Population (P): patients with massive bone resorption horizontally and vertically, severe bone loss around teeth, periodontal disease or traumatic extraction in partially edentulous maxillary anterior region requiring implant insertion.

Intervention (I): simultaneous implant placement with ridge augmentation using computer guided surgical templates with PRF.

Comparator (C): Free hand simultaneous implant placement with ridge augmentation.

Outcome (O): Patient esthetic satisfaction - Augmentation and implant insertion accuracy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with insufficient alveolar ridge or severe alveolar bone resorption horizontally and vertically in partially edentulous maxillary anterior region.
2. Medically free patients in order to be a confounding factor on the final results.
3. Highly motivated patients.
4. Good oral hygiene.
5. Patients physically able to tolerate surgical and restorative procedures.

Exclusion Criteria:

1. Young patients (incomplete bone growth).
2. Patients with any systemic disease that could affect bone healing.
3. Patients allergic to local anaesthetic agent.
4. Pregnant or lactating females.
5. Presence of any pathosis in the area.
6. history of oral radiotherapy.
7. history of prolonged steroid use.
8. Psychological disorders.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction regarding esthetic results. | 5 month
  outcome will be measured using questionnaire

SECONDARY OUTCOMES:
Accuracy of computer guided surgical templates in comparison with 3D virtual planning. | immediately after procedure
  Comparing the results on the patient with the design made by the surgical software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Evaluation of The Comparative Effectiveness of Computer Guided Surgical stents in Anterior Ridge Defects with Bone Ring Graft and PRF

REFERENCES:
- [Background] Omara M, Abdelwahed N, Ahmed M, Hindy M. Simultaneous implant placement with ridge augmentation using an autogenous bone ring transplant. Int J Oral Maxillofac Surg. 2016 Apr;45(4):535-44. doi: 10.1016/j.ijom.2015.11.001. Epub 2015 Nov 28. PMID 26644216